CLINICAL TRIAL: NCT01137500
Title: Ultrasonic Assessment of Changes in Aortic Diameter During Laparoscopic Surgery
Brief Title: Changes in Aortic Diameter During Laparoscopic Surgery
Status: Withdrawn | Type: Observational
Why Stopped: host site logistical problems
Sponsor: Royal Surrey County Hospital NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Dr Matthew Dickinson, Anaesthetist, Royal Surrey County Hospital NHS Foundation Trust
Other Study IDs: RSCHanaes001
Record Dates: First submitted 2010-06-03; First posted 2010-06-04 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Abdominal Aortic Diameter During Laparoscopic Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Various haemodynamic changes are observed during laparoscopic surgery, relating to insufflation of CO2 & patient position. Cardiac output calculations using oesophageal doppler monitoring are based on the assumption that the aortic diameter is fixed. This study aims to measure the aortic diameter at preset times during surgery using ultrasound to discover if the diameter remains the same, and hence if the assumptions made by the oesophageal monitor are reliable. Assessing the aortic diameter involves a noninvasive ultrasound measurement taken in patients electively having laparoscopic procedures at the Royal Surrey County Hospital.

DETAILED DESCRIPTION:
Purpose and design:This study aims to measure the aortic diameter at preset times during surgery using ultrasound to discover if the diameter remains the same, and hence if the assumptions made by the oesophageal monitor are reliable. Assessing the aortic diameter involves a noninvasive ultrasound measurement taken in patients electively having laparoscopic procedures at the Royal Surrey County Hospital.

Recruitment: Patients undergoing elective laparoscopic procedures at the Royal Surrey County Hospital. Recruitment done by Dr M Dickinson or Dr M Scott (COnsultant Anaesthetists). No therapeutic promises are to be made as this is purely an observational study.

Inclusion / exclusion: Patient refusal, Surgical refusal, Conversion to an open procedure.

Consent: Informed consent will be gained from each participant.

Risks, burdens and benefits: This is an observational study using a non invasive technique in patients undergoing elective surgery. There is very little in the way of risks, burdens and benefits to the patient.

Confidentiality: Caldicott principles will be adhered to.

Conflict of interest: None.

Use of tissue samples in future research: None.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients undergoing elective laparoscopic surgery at the Royal Surrey County Hospital

Exclusion Criteria:

* Patient refusal
* Surgical refusal
* Conversion to an open procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective laparoscopic procedures at the Royal Surrey County Hospital. Recruitment done by Dr M Dickinson or Dr M Scott (COnsultant Anaesthetists). No therapeutic promises are to be made as this is purely an observational study
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-08-01 (Actual); Primary Completion 2010-08-02 (Actual); Study Completion 2010-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew C Dickinson, MB BS, Principal Investigator — Royal Surrey County Hospital NHS Foundation Trust; Mike Scott, MB BS, Study Director — Royal Surrey County Hospital NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: No